CLINICAL TRIAL: NCT07167667
Title: Investigation of the Effects of Two Different Physiotherapy Modalities on Median Nerve Thickness, Electrophysiological Activity, Pain Intensity and Quality of Life in Patients With Carpal Tunnel Syndrome - An Observational Study
Brief Title: Median Nerve Thickness of the Carpal Tunnel Syndrome After Two Different Physiotherapy Modalities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emre Şenocak (Other)
Responsible Party: Sponsor-Investigator, Emre Şenocak, Assistant Professor, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/145
Record Dates: First submitted 2025-06-11; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Median Nerve Thickness; Ultrasound; Electromyograpy; Physiotherapy; ESWT; Paraffin
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paraffin (Experimental)
  Interventions: Other: Paraffin Bath
- ESWT (Experimental)
  Interventions: Other: Extracorporeal Shock Wave Therapy

INTERVENTIONS:
Other: Paraffin Bath — Patients' hands will be dipped into the paraffin bath 8-10 times.
  Arms: Paraffin
Other: Extracorporeal Shock Wave Therapy — The patients will be treated with a sound wave pulse frequency of 15 Hz, an intensity of 1.5 bar, and a total number of pulses of 2000 for one session.
  Arms: ESWT

SUMMARY:
The study plans to include a total of 60 patients diagnosed with carpal tunnel syndrome. Patients will be divided into two groups according to the treatment they receive. One group will receive only paraffin treatment, while the other group will receive only ESWT treatment. ESWT will be applied for a total of 5 sessions. Paraffin will be applied for a total of 10 sessions. As assessment tools;

* Measurement of median nerve thickness with ultrasound
* Electromyography
* Visual Analog Scale
* Short Form-36

Evaluations will be made twice by a specialist physician before and after the treatments.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 30-60 who have been diagnosed with CTS by a specialist physician according to international criteria (Those between Stages 1-3),
* Those who have complaints of numbness, tingling, and pain in the first three fingers and half of the fourth finger,
* Phalen Test and Tinel sign or Durkan Test being positive
* Patients who will receive 5 sessions of ESWT application prescribed by a Physical Medicine and Rehabilitation Specialist Physician (for the ESWT group)
* Patients who have been recommended 10 sessions of Paraffin application by a Physical Medicine and Rehabilitation Specialist Physician (for the Paraffin group)

Exclusion Criteria:

* Presence of atrophy in the thenar muscles,
* Insufficient sensory and motor response in the median nerve,
* History of hand and/or wrist injury or surgery,
* Those with cervical stenosis, cervical spondylosis, or cervical radiculopathy,
* Corticosteroids in the carpal tunnel area within the last six months those who have had an injection,
* Pregnancy or diabetes, renal failure, rheumatoid arthritis or hypothyroidism

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-10-25 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
Median Nerve Thickness | Baseline
  Median nerve thickness will be measured by ultrasound
Median Nerve Thickness | 5 days later for the first ESWT intervention and 10 days later for the first Paraffin Intervention
  Median nerve thickness will be measured by ultrasound

SECONDARY OUTCOMES:
Electromyography | Baseline
  EMG will be used to diagnose carpal tunnel.
Visual Analog Scale | Baseline
  It will be used to assess pain intensity.
Visual Analog Scale | 5 days later for the first ESWT intervention and 10 days later for the first Paraffin Intervention
  It will be used to assess pain intensity.
Short Form-36 | Baseline
  It will be used to evaluate patients' quality of life.
Short Form-36 | 5 days later for the first ESWT intervention and 10 days later for the first Paraffin Intervention
  It will be used to evaluate patients' quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Baltalimani Metin Sabanci Bone Diseases Training and Research Hospita, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No